CLINICAL TRIAL: NCT02554903
Title: A Prospective, Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety of Macitentan in Patients With Pulmonary Hypertension After Left Ventricular Assist Device Implantation
Brief Title: Clinical Study to Assess the Efficacy and Safety of Macitentan in Patients With Pulmonary Hypertension After Left Ventricular Assist Device Implantation
Acronym: SOPRANO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC-055-205
Record Dates: First submitted 2015-09-08; First posted 2015-09-18 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Hypertension
Keywords: LVAD
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — macitentan; Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Macitentan 10 mg po (Experimental): Approximately 78 adult subjects with PH post-LVAD implantation will be randomized (1:1) to receive either macitentan 10 mg, or matching placebo, once daily orally.
  Interventions: Drug: Macitentan 10mg
- Placebo sugar pill (Placebo Comparator): Approximately 78 adult subjects with PH post-LVAD implantation will be randomized (1:1) to receive either macitentan 10 mg, or matching placebo, once daily orally.
  Interventions: Drug: Placebo sugar pill

INTERVENTIONS:
Drug: Macitentan 10mg — 2 groups, randomized in a 1:1 ratio by an Interactive Voice/Web Randomization System to macitentan 10 mg or placebo
  Other Names: Active drug
  Arms: Macitentan 10 mg po
Drug: Placebo sugar pill — 2 groups, randomized in a 1:1 ratio by an Interactive Voice/Web Randomization System to macitentan 10 mg or placebo
  Other Names: placebo comparator
  Arms: Placebo sugar pill

SUMMARY:
STUDY OBJECTIVES Primary objective To evaluate the effect of macitentan 10 mg on pulmonary vascular resistance (PVR) as compared to placebo in subjects with pulmonary hypertension (PH) after left ventricular assist device (LVAD) implantation.

Secondary objectives To evaluate the effect of macitentan 10 mg as compared to placebo on cardio-pulmonary hemodynamics and disease severity in subjects with PH after LVAD implantation.

To evaluate the safety and tolerability of macitentan 10 mg in subjects with PH after LVAD implantation.

Exploratory objectives To explore the potential effect of macitentan 10 mg as compared to placebo on right ventricular function in subjects with PH after LVAD implantation.

To explore the potential effect of macitentan 10 mg as compared to placebo on selected clinical events in subjects with PH after LVAD implantation.

To explore the potential effect of macitentan 10 mg as compared to placebo on renal function as measured by glomerular filtration rate (GFR) in subjects with PH after LVAD implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent prior to initiation of any study-mandated procedure.
2. Males or females ≥ 18 years of age.
3. Surgical implantation of LVAD within 90 days prior to Randomization.
4. Hemodynamic evidence of PH on Baseline right heart catheterization (RHC) by the thermodilution method. Baseline RHC is defined as the last hemodynamic measurements after LVAD implantation and prior to the first dose of study treatment. PH is defined as:

   1. Mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg and
   2. Pulmonary artery wedge pressure (PAWP) ≤ 18 mmHg and
   3. PVR > 3 Wood units.
5. Stabilization of the patient for 48 h prior to the Baseline RHC, defined as:

   1. No LVAD pump speed/flow rate changes and
   2. Stable dose of oral diuretics and
   3. No intravenous (i.v.) inotropes or vasopressors and
   4. Patient able to ambulate.
6. A woman of childbearing potential is eligible only if she has:

   1. A negative serum pregnancy test result during the Screening period (Visit 1) and Randomization (Visit 2) and
   2. Agreement to undertake monthly serum pregnancy tests during the study and up to 30 days after study treatment discontinuation and
   3. Agreement to use one of the methods of contraception / follow the contraception scheme described in Section 4.5 from Screening and up to at least 30 days after study treatment discontinuation.
7. Patient must be randomized within 14 days of Baseline RHC.

Exclusion Criteria:

1. Documented severe obstructive lung disease defined as: forced expiratory volume in 1 second / forced vital capacity (FEV1/FVC) < 0.7 associated with FEV1 < 50% of predicted value after bronchodilator administration.
2. Documented moderate to severe restrictive lung disease defined as: total lung capacity < 60% of predicted value.
3. Documented pulmonary veno-occlusive disease.
4. Patients undergoing dialysis.
5. Hemoglobin < 8.5 g/dL at Randomization.
6. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 × the upper limit of normal (ULN) at Randomization.
7. Severe hepatic impairment, e.g., Child-Pugh Class C liver disease.
8. Body weight < 40 kg at Randomization.
9. Doppler mean blood pressure < 65 mmHg at Randomization.
10. GFR < 30 mL/min at Randomization.
11. Pregnant, planning to become pregnant during the study period, or breastfeeding.
12. Treatment with endothelin receptor antagonists (ERAs), phosphodiesterase-5 (PDE5) inhibitors, i.v., subcutaneous (s.c.), or oral prostanoids, or guanylate cyclase stimulators within 7 days prior to Baseline RHC or study treatment initiation.
13. Treatment with inhaled prostanoids (e.g., iloprost, epoprostenol) or nitric oxide within 24 h prior to Baseline RHC or study treatment initiation.
14. Treatment with strong inducers of cytochrome P450 isozyme 3A4 (CYP3A4) within 28 days prior to study treatment initiation (e.g., carbamazepine, rifampicin, rifabutin, phenytoin and St. John's Wort).
15. Treatment with strong inhibitors of CYP3A4 within 28 days prior to study treatment initiation (e.g., ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, nefazodone, ritonavir, saquinavir, boceprevir, telaprevir, iopinavir, fosamprenavir, darunavir, tipranavir, atazanavir, nelfinavir, amprenavir, and idinavir).
16. Treatment with another investigational drug (planned, or taken) within 28 days prior to study treatment initiation.
17. Known hypersensitivity to ERAs, or to any of the study treatment excipients.
18. Any condition that prevents compliance with the protocol or adherence to therapy.
19. Known concomitant life-threatening disease with a life expectancy < 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rocco, Study Director — Actelion
Locations (50):
- United States (50):
  - #125_Mayo Clinic Arizona, Phoenix, Arizona
  - #144_University of Arizona, Tucson, Arizona
  - #106_Cedars-Sinai Medical Center, Beverly Hills, California
  - #154_University of California San Diego, La Jolla, California
  - #110_Sutter Heart Institute, Sacramento, California
  - #132_University of California San Francisco, San Francisco, California
  - #123_MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - #126_Florida Hospital, Orlando, Florida
  - #135_University of Chicago Medical Center, Chicago, Illinois
  - #113_Advocate Christ Medical Center, Oak Lawn, Illinois
  - #108_Indiana University Health Physicians Cardiology, Indianapolis, Indiana
  - #112_St. Vincent Medical Group, Inc, Indianapolis, Indiana
  - #120_University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - #117_University of Louisville, Louisville, Kentucky
  - #105_Ochsner Medical Center, New Orleans, Louisiana
  - #129_John Hopkins University Medical Center, Baltimore, Maryland
  - #143_Tufts Medical Center, Boston, Massachusetts
  - #138_Massachusetts General Hospital, Boston, Massachusetts
  - #119_Brigham and Women's Hospital, Boston, Massachusetts
  - #115_Henry Ford Hospital, Detroit, Michigan
  - #102_Mayo Clinic, Rochester, Minnesota
  - #150_Saint Luke's Hospital, Kansas City, Missouri
  - #104_Washington University School of Medicine, St Louis, Missouri
  - #131_University of Nebraska Medical Center, Omaha, Nebraska
  - #103_Weill Cornell Medical College, New York, New York
  - #139_Icahn School of Medicine at Mount Sinai, New York, New York
  - #133_Montefiore Medical Center, The Bronx, New York
  - #147_Westchester Medical Center, Valhalla, New York
  - #148_University of Cincinnati Medical Center, Cincinnati, Ohio
  - #153_Cleveland Clinic, Cleveland, Ohio
  - #101_The Ohio State University Wexner Medical Center, Columbus, Ohio
  - #145_The University of Toledo Medical Center, Toledo, Ohio
  - #121_Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - #142_Penn State Heart and Vascular Institute, Hershey, Pennsylvania
  - #140_Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - #134_Allegheny General Hospital, Pittsburgh, Pennsylvania
  - #130_University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - #141_Palmetto Health / Palmetto Heart, Columbia, South Carolina
  - #151_Stern Cardiovascular Foundation, Memphis, Tennessee
  - #146_Vanderbilt University Medical Center, Nashville, Tennessee
  - #149_Seton Heart Institute, Austin, Texas
  - #136_Baylor Health - Baylor University Medical Center, Dallas, Texas
  - #107_Houston Methodist Hospital, Houston, Texas
  - #122_Advanced Heart Failure Clinic - HCM, San Antonio, Texas
  - #127_The University of Utah, Salt Lake City, Utah
  - #114_University of Virginia, Charlottesville, Virginia
  - #111_Inova Fairfax Hospital, Falls Church, Virginia
  - #116_Virginia Commonwealth University (VCU) Medical Center, Richmond, Virginia
  - #155_University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Frantz RP, Desai SS, Ewald G, Franco V, Hage A, Horn EM, LaRue SJ, Mathier MA, Mandras S, Park MH, Ravichandran AK, Schilling JD, Wang IW, Zolty R, Rendon GG, Rocco MA, Selej M, Zhao C, Rame JE. SOPRANO: Macitentan in patients with pulmonary hypertension following left ventricular assist device implantation. Pulm Circ. 2024 Dec 4;14(4):e12446. doi: 10.1002/pul2.12446. eCollection 2024 Oct. PMID 39635465

RESULTS

PARTICIPANT FLOW:
Groups:
- Macitentan 10 Milligrams (mg): Participants (with pulmonary hypertension [PH] after a left ventricular assist device [LVAD] implantation) received macitentan 10 mg orally once daily up to Week 12.
- Placebo: Participants (with PH after LVAD implantation) received matching placebo orally once daily up to Week 12.
Period: Overall Study
Arm/Group | Macitentan 10 Milligrams (mg) | Placebo
Started | 28 | 29
Completed | 24 | 24
Not Completed | 4 | 5
Not completed — Death | 1 | 1
Not completed — Physician Decision | 2 | 2
Not completed — Heart Transplant | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Macitentan 10 Milligrams (mg) | Placebo | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (8.21) | 58.2 (6.98) | 57.4 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 22 | 23 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Black or African American | 8 | 11 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 16 | 18 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
  Other | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Vascular Resistance (PVR) Ratio of Week 12 to Baseline
Description: PVR ratio equals to Week 12 PVR / Baseline PVR. PVR represents the resistance against which the right ventricle needs to pump. PVR was calculated using the following formula: mean pulmonary arterial pressure (mPAP) - pulmonary artery wedge pressure (PAWP)/cardiac output (CO); where mPAP and PAWP were measured at end-expiration and CO was measured in triplicate using the thermodilution method.
Time Frame: Baseline to Week 12
Population: The Full Analysis Set (FAS) included all participants randomized. Here 'N' (number of participants analyzed) included all participants who were evaluable for this outcome measure. Imputation for missing PAWP value was done using mPAP and CO or with left ventricular end diastolic pressure (LVEDP) values of same visit (if available).
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Placebo: Participants (with PH after a LVAD implantation) received matching placebo orally once daily up to Week 12.
Arm/Group | Macitentan 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 27 | 28
Ratio | 0.585 (0.2280) | 0.757 (0.2578)
Statistical Analysis 1: Comparison: Macitentan 10 Milligrams (mg) vs Placebo; Test type: Superiority; p = 0.0158, ANCOVA; Geometric Mean Ratio = 0.7393, 95% CI 2-sided [0.5798 to 0.9426]

2. Secondary Outcome: Change From Baseline to Week 12 in Mean Right Atrial Pressure (mRAP)
Description: mRAP was collected in the eCRF (electronic case record form). Right atrial pressure (RAP) is the blood pressure in the right atrium of the heart. Change from baseline to Week 12 in mRAP was measured at rest and no correction for multiple testing was applied.
Time Frame: Baseline to Week 12
Population: The FAS included all participants randomized. Here 'N' (number of participants analyzed) included all participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Groups:
- Macitentan 10 Milligrams (mg): Participants (with PH after a LVAD implantation) received macitentan 10 mg orally once daily up to Week 12.
Arm/Group | Macitentan 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 25 | 25
millimeters of mercury (mmHg) | 0.8 (5.49) | -1.4 (4.71)

3. Secondary Outcome: Change From Baseline to Week 12 in Mean Pulmonary Arterial Pressure (mPAP)
Description: mPAP was collected in the eCRF. The pulmonary artery pressure is a measure of the blood pressure found in the main pulmonary artery. Change from baseline to Week 12 in mPAP was measured at rest and no correction for multiple testing was applied.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Macitentan 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 25 | 25
mmHg | -3.84 (8.821) | -3.86 (7.982)

4. Secondary Outcome: Change From Baseline to Week 12 in Pulmonary Arterial Wedge Pressure (PAWP)
Description: PAWP was collected in the eCRF. PAWP is pressure within the pulmonary arterial system when the catheter tip is 'wedged' in the tapering branch of one of the pulmonary arteries. Change from baseline to Week 12 in PAWP was measured at rest and no correction for multiple testing was applied.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Macitentan 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 25 | 25
mmHg | 4.0 (7.86) | 1.0 (4.93)

5. Secondary Outcome: Change From Baseline to Week 12 in Cardiac Index (CI)
Description: CI was calculated as Cardiac Output (CO)/body surface area (BSA), where CO is Thermodilution Cardiac Output (Liters per minute [L/min]) and BSA (m^2) equals to 0.007184*weight^0.425 (kilograms)*height^0.725 (centimeter). CI was represented in liters per minute per square meter (L/min/m^2). Change from baseline to Week 12 in CI was measured at rest and no correction for multiple testing was applied.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Macitentan 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 24 | 25
L/min/m^2 | 0.093 (0.4680) | 0.041 (0.4576)

6. Secondary Outcome: Change From Baseline to Week 12 in Total Pulmonary Resistance (TPR)
Description: TPR was calculated as mPAP/CO where mPAP is mean pulmonary arterial pressure and CO is cardiac output. Change from baseline to Week 12 in TPR was calculated at rest and no correction for multiple testing was applied.
Time Frame: Baseline to Week 12
Population: The FAS included all participants randomized. Here 'N' (number of participants analyzed) includes all participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Wood Unit
Arm/Group | Macitentan 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 24 | 25
Wood Unit | -1.399 (2.2515) | -0.993 (2.2596)

7. Secondary Outcome: Change From Baseline to Week 12 in Mixed Venous Oxygen Saturation (SvO2)
Description: Mixed venous oxygen saturation measures the end result of oxygen consumption and delivery. Change from baseline to Week 12 in SvO2 was reported and measured at rest and no correction for multiple testing was applied.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of SvO2
Arm/Group | Macitentan 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 25 | 25
Percentage of SvO2 | 4.260 (17.1523) | 4.100 (8.5202)

8. Secondary Outcome: Change From Baseline to Week 12 in N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP) Levels
Description: NT-proBNP levels in the blood are used for diagnosis of acute congestive heart failure (CHF) and may be useful to establish prognosis in heart failure.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanograms/Liter (ng/L)
Arm/Group | Macitentan 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 22 | 25
nanograms/Liter (ng/L) | 1325.68 (1214.719) | 1573.44 (2327.632)

9. Secondary Outcome: Change From Baseline to Week 12 in Participants World Health Organization (WHO) Functional Class (FC)
Description: WHO FC is a classification which reflects disease severity based on symptoms. WHO Functional Classification of pulmonary hypertension comprises of Class I (participants with pulmonary hypertension but without resulting limitation of physical activity), II (participants with pulmonary hypertension resulting in slight limitation of physical activity), III (participants with pulmonary hypertension resulting in marked limitation of physical activity) and IV (participants with pulmonary hypertension with inability to carry out any physical activity without symptoms). Change from baseline in WHO FC was reported. WHO FC was categorized as worsening (change greater than [>] 0); improvement (change less than [<] 0); or no change (change equals to [=] 0).
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 25 | 25
Participants
  Worsening | 2 | 2
  No change | 13 | 15
  Improvement | 10 | 8

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Description: The safety analysis included all participants who received at least one dose of study drug.
Arm/Group | Macitentan 10 Milligrams (mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 1/28 | 2/29
Serious Adverse Events (participants affected / at risk) | 16/28 | 16/29
Other Adverse Events (participants affected / at risk) | 24/28 | 24/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 10 Milligrams (mg) (N=28) | Placebo (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Leukaemoid Reaction (Blood and lymphatic system disorders) | 0 | 1
Atrial Flutter (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0
Cardiac Failure Acute (Cardiac disorders) | 1 | 1
Right Ventricular Failure (Cardiac disorders) | 2 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Complication Associated with Device (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Peripheral Swelling (General disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Enterococcal Bacteraemia (Infections and infestations) | 1 | 0
Groin Abscess (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 2 | 0
Streptococcal Infection (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Anticoagulation Drug Level below Therapeutic (Investigations) | 3 | 4
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 1 | 0
International Normalised Ratio Increased (Investigations) | 1 | 1
Left Ventricular End-Diastolic Pressure Increased (Investigations) | 1 | 0
Liver Function Test Increased (Investigations) | 1 | 0
Troponin Increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Fluid Retention (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Chest Wall Haematoma (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Haemorrhagic Stroke (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Reversible Ischaemic Neurological Deficit (Nervous system disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 10 Milligrams (mg) (N=28) | Placebo (N=29)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Atrial Flutter (Cardiac disorders) | 1 | 1
Cardiogenic Shock (Cardiac disorders) | 1 | 0
Cardiorenal Syndrome (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Systolic Dysfunction (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 1
Vision Blurred (Eye disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Gingival Bleeding (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 4
Asthenia (General disorders) | 1 | 0
Catheter Site Haemorrhage (General disorders) | 0 | 2
Chest Discomfort (General disorders) | 1 | 0
Complication Associated with Device (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 1
Feeling Abnormal (General disorders) | 0 | 1
Impaired Healing (General disorders) | 1 | 0
Medical Device Site Discharge (General disorders) | 0 | 1
Medical Device Site Erythema (General disorders) | 0 | 1
Medical Device Site Rash (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 4 | 1
Pain (General disorders) | 0 | 1
Peripheral Swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Candida Infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Medical Device Site Infection (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2
Ophthalmic Herpes Simplex (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 3
Fractured Sacrum (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Anticoagulation Drug Level above Therapeutic (Investigations) | 0 | 1
Anticoagulation Drug Level below Therapeutic (Investigations) | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 2 | 2
Blood Glucose Increased (Investigations) | 0 | 1
Blood Potassium Decreased (Investigations) | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 2
Blood Sodium Decreased (Investigations) | 1 | 0
Blood Triglycerides Increased (Investigations) | 1 | 0
Blood Urea Increased (Investigations) | 2 | 2
Blood Uric Acid Increased (Investigations) | 2 | 0
Body Temperature Increased (Investigations) | 0 | 1
Cystatin C Increased (Investigations) | 3 | 0
Echocardiogram Abnormal (Investigations) | 0 | 1
Ejection Fraction Decreased (Investigations) | 1 | 0
Electrocardiogram St Segment Elevation (Investigations) | 1 | 0
Haematocrit Decreased (Investigations) | 1 | 0
Haemoglobin Abnormal (Investigations) | 1 | 0
Haemoglobin Decreased (Investigations) | 1 | 0
Heart Rate Irregular (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 1
International Normalised Ratio Increased (Investigations) | 0 | 1
N-Terminal Prohormone Brain Natriuretic Peptide Increased (Investigations) | 4 | 4
Platelet Count Decreased (Investigations) | 0 | 1
Protein Total Decreased (Investigations) | 1 | 0
Smear Cervix Abnormal (Investigations) | 1 | 0
Troponin Increased (Investigations) | 1 | 1
Venous Pressure Jugular Increased (Investigations) | 0 | 1
Weight Decreased (Investigations) | 0 | 1
Weight Increased (Investigations) | 2 | 0
White Blood Cell Count Increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Fluid Overload (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 7
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Lumbosacral Radiculopathy (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Breast Tenderness (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea Paroxysmal Nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Chronic Pigmented Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypersensitivity Vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Palpable Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Tightness (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 2 | 1
Orthostatic Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
A limitation of this study was its slow enrollment and a final sample size that was less than the predefined target.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT02554903/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT02554903/SAP_001.pdf